CLINICAL TRIAL: NCT02850900
Title: Oral Psoriasis Treatment Adherence and Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00035938
Record Dates: First submitted 2016-05-05; First posted 2016-08-01 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet Survey (Experimental): Subject will receive an electronic survey weekly to complete
  Interventions: Behavioral: Internet Survey
- No Survey (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Internet Survey — Weekly survey will be emailed, subjects should complete them
  Arms: Internet Survey

SUMMARY:
Response to psoriasis treatment is variable in large part because of poor adherence treatments. Studies using electronic monitors have assessed adherence to topical and injectable psoriasis treatments and to biologics, yielding critically important insights. Adherence to oral psoriasis treatments is not as well characterized but is also critical, as the therapeutic windows for these treatments are narrower than for other psoriasis treatment options.

The proposed study will assess patients' adherence to oral psoriasis treatment (primarily methotrexate) and will also collect pilot data on an intervention to improve adherence. The primary hypothesis of the investigators study is that adherence to oral psoriasis treatment is poor and that a reporting intervention may improve adherence to oral psoriasis treatment. In the investigator-blinded, 6-month prospective study, patients will be randomized to standard-of-care treatment or standard-of-care supplemented with the weekly online reporting intervention. Adherence will be assessed using electronic monitors. This randomized trial will permit the investigators to determine adherence to oral psoriasis treatment, assess the relationship between adherence and psoriasis outcomes, identify factors that are associated with adherence to oral psoriasis treatment (including physician trust, confidence in the treatment plan, and depression), and obtain preliminary data on the impact of an Internet-reporting measure on patients' adherence to oral psoriasis treatment

.

DETAILED DESCRIPTION:
Psoriasis is a common, chronic inflammatory disease that has a major impact on patients' quality of life. Patients' response to treatment is variable. Poor adherence to topical, oral and biologic psoriasis treatments is common and may account for poor responses.1, 2 Many psoriasis patients do not even fill their prescriptions.3 Electronic monitoring of adherence provides the most detailed and accurate way to assess adherence. While studies using electronic monitors have assessed adherence to topical psoriasis treatments and to biologics, adherence to oral psoriasis treatments is not as well characterized. Understanding adherence to oral psoriasis treatments is critical, as the therapeutic windows for these treatments are narrower than for other psoriasis treatment options, making adherence to recommended dosing all the more critical.

Developing methods to improve psoriasis patients' adherence has the potential to provide an immediate, practical means to improve patients' treatment outcomes. Return visits improve patients' use of medication & treatment outcomes but are not practical and add additional costs to the patient and medical system. Having patients report on their treatment experience without an office visit offers promise for improving adherence but has not been tested in a psoriasis population.

The primary hypothesis of the investigators study is that adherence to oral psoriasis treatment is poor and that a reporting intervention may improve adherence to oral psoriasis treatment.

The Specific Aims of this study are:

1. To determine adherence to oral psoriasis treatments (methotrexate) with electronic monitors.
2. To assess the relationship between adherence and psoriasis outcomes (measured by body surface area [BSA], Physician Global Assessment [PGA] and [BSA]x[PGA]).
3. To identify factors that are associated with adherence to oral psoriasis treatment, including physician trust, confidence in the treatment plan, and depression which will be measured with the Wake Forest University Physician Trust Scale (WFUPTS),4-6 the Treatment Satisfaction Questionnaire for Medication (TSQM),7 and the Hamilton Depression Rating Scale (HAM-D).
4. To test obtain preliminary data on the impact of an Internet-reporting measure on patients' adherence to oral psoriasis treatment.

The investigators propose an investigator-blinded, 6-month prospective study of 40 patients aged 12 and older who have been prescribed oral psoriasis treatment. Adherence will be assessed using Medication Event Monitoring System (MEMS®) caps, electronic monitors affixed to the medication containers. Investigators and subjects will be blinded to the adherence data until the final (Month 6) treatment visit.

This study is of high significance, providing critically important information on how patients use oral psoriasis treatments, as well as a foundation to develop and implement intervention trials to improve adherence and outcomes in patients treated with oral psoriasis treatments. Innovations in this study include seeking to change the paradigm of the investigators understanding of the role of adherence in oral psoriasis treatment, including effects on treatment failures and side effects, developing a new understanding of the roles of physician and medication trust in adherence, and potentially changing the timing and methods of clinical assessments in psoriasis (and other) patients in light of the effects of the timing and methods of clinical assessments on treatment adherence and outcomes. The use of objective electronic adherence monitors and well-validated assessment tools adds strength to the approach of this study; another strength of the approach is careful attention to research ethics of adherence monitoring. The environment of this study is particularly strong, with facilities for and extensive experience in all aspects of adherence monitoring research.

The overall goal of this study is to better understand and improve adherence behaviors in patients with psoriasis, a common, chronic, relapsing, inflammatory disease. Psoriasis reduces patients' quality of life, yet patients with psoriasis, as with other chronic diseases, frequently misuse medicine, impairing effectiveness of prescribed therapies (when underused) and increasing the risks of treatment (when overused or mistimed).8 Poor adherence to treatment can be misconstrued as poor response, which can lead to unnecessary treatment escalation resulting in exposing patients to more toxic or costly medications.9 In many cases, non-adherence, rather than non-response, is the underlying precursor of treatment failure.10, 11

Adherence issues with oral psoriasis treatment are largely unexplored and are of critical importance. Oral methotrexate is widely used (encouraged by payors), yet it is risky, with a more narrow therapeutic window than biologics. Other oral agents approved for psoriasis include cyclosporine (with a risk of renal disease) and apremilast (which is associated with gastrointestinal tolerability issues). While large database studies find that oral psoriasis treatment is underused, the variation in use of oral psoriasis treatments among patients is critically important and has not been defined.

Traditional methods for measuring medical adherence tend to be unreliable. Assessment methods such as patient interviews, questionnaires, surveys, and diaries deliver inconsistent data that depend upon the patient's willingness to accurately record medication use and ability to remember what they did. Electronic monitoring devices offer an effective means for objective adherence monitoring. Medication Event Monitoring System caps (MEMS®, AARDEX Corp., Fremont, CA) include microprocessors in the bottle cap of a standard medication bottle that record each time and date the bottle is opened and the interval since the last bottle opening.12

The availability of accurate electronic adherence measurement provides a foundation to study novel ways to improve adherence. In several studies of psoriasis and other inflammatory skin diseases, a clear pattern of improved adherence around the time of office visits is evident. The tendency for patients to be more adherent around the time of office visits may be a form of a more general tendency to be adherent when interacting with the healthcare system to assess their treatment outcomes, a form of "white coat compliance" or Hawthorne effect. A pilot study of adolescents with acne vulgaris tested whether adherence to topical benzoyl peroxide could be improved by weekly online-reporting of their treatment experience.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female 12 years or older of age with a diagnosis of psoriasis who is prescribed methotrexate by a dermatologist will be eligible for participation.
* Greater than 10% of body surface involvement for psoriasis.
* Subject is capable of understanding and willing to provide a signed and dated written voluntary informed consent before any protocol specific procedures are performed.
* The subject is able to complete the study and comply with study instructions, including attending all study visits.

Exclusion Criteria:

* Individuals younger than 12 years of age.
* Known allergy or sensitivity to methotrexate.
* Inability to complete all study-related visits, or inability to complete the Internet survey due to inadequate Internet access.
* Introduction of any other prescription medication, topical or systemic, for psoriasis while participating in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed oral Methotrexate treatment | 6 months
  Determined by intervention of weekly internet survey compared to no survey
Patterns of Misuse | 6 months
  Self-report of not taking the medication as prescribed;
Psoriasis severity outcomes | 6 months
  The relationship between body surface area, Physician Global Assessment outcomes will be assessed.

SECONDARY OUTCOMES:
Relationship to Adherence | 6 months
  It will be explored using physician trust scale, a validated tool.
Relationship to Satisfaction | 6 months
  It will be explored using the treatment and satisfaction survey, a validated survey.

CONTACTS AND LOCATIONS:
Overall Officials: William H Huang, MD, Principal Investigator — Wake Forest
Locations (1):
- Wake Forest University School of Medicine - Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
will determine at later date

REFERENCES:
- [Background] Richards HL, Fortune DG, O'Sullivan TM, Main CJ, Griffiths CE. Patients with psoriasis and their compliance with medication. J Am Acad Dermatol. 1999 Oct;41(4):581-3. PMID 10495380
- [Background] Carroll CL, Feldman SR, Camacho FT, Balkrishnan R. Better medication adherence results in greater improvement in severity of psoriasis. Br J Dermatol. 2004 Oct;151(4):895-7. doi: 10.1111/j.1365-2133.2004.06174.x. PMID 15491434
- [Background] Storm A, Andersen SE, Benfeldt E, Serup J. One in 3 prescriptions are never redeemed: primary nonadherence in an outpatient clinic. J Am Acad Dermatol. 2008 Jul;59(1):27-33. doi: 10.1016/j.jaad.2008.03.045. Epub 2008 May 7. PMID 18467003
- [Background] Balkrishnan R, Dugan E, Camacho FT, Hall MA. Trust and satisfaction with physicians, insurers, and the medical profession. Med Care. 2003 Sep;41(9):1058-64. doi: 10.1097/01.MLR.0000083743.15238.9F. PMID 12972845
- [Background] Hall MA, Dugan E, Zheng B, Mishra AK. Trust in physicians and medical institutions: what is it, can it be measured, and does it matter? Milbank Q. 2001;79(4):613-39, v. doi: 10.1111/1468-0009.00223. PMID 11789119
- [Background] Hall MA, Zheng B, Dugan E, Camacho F, Kidd KE, Mishra A, Balkrishnan R. Measuring patients' trust in their primary care providers. Med Care Res Rev. 2002 Sep;59(3):293-318. doi: 10.1177/1077558702059003004. PMID 12205830
- [Background] Atkinson MJ, Sinha A, Hass SL, Colman SS, Kumar RN, Brod M, Rowland CR. Validation of a general measure of treatment satisfaction, the Treatment Satisfaction Questionnaire for Medication (TSQM), using a national panel study of chronic disease. Health Qual Life Outcomes. 2004 Feb 26;2:12. doi: 10.1186/1477-7525-2-12. PMID 14987333
- [Background] Murphy J, Coster G. Issues in patient compliance. Drugs. 1997 Dec;54(6):797-800. doi: 10.2165/00003495-199754060-00002. PMID 9421690
- [Background] Frances C, Cosnes A, Duhaut P, Zahr N, Soutou B, Ingen-Housz-Oro S, Bessis D, Chevrant-Breton J, Cordel N, Lipsker D, Costedoat-Chalumeau N. Low blood concentration of hydroxychloroquine in patients with refractory cutaneous lupus erythematosus: a French multicenter prospective study. Arch Dermatol. 2012 Apr;148(4):479-84. doi: 10.1001/archdermatol.2011.2558. PMID 22508872
- [Background] Eisen SA, Woodward RS, Miller D, Spitznagel E, Windham CA. The effect of medication compliance on the control of hypertension. J Gen Intern Med. 1987 Sep-Oct;2(5):298-305. doi: 10.1007/BF02596162. PMID 3655955
- [Background] Paterson DL, Swindells S, Mohr J, Brester M, Vergis EN, Squier C, Wagener MM, Singh N. Adherence to protease inhibitor therapy and outcomes in patients with HIV infection. Ann Intern Med. 2000 Jul 4;133(1):21-30. doi: 10.7326/0003-4819-133-1-200007040-00004. PMID 10877736
- [Background] Urquhart J. The electronic medication event monitor. Lessons for pharmacotherapy. Clin Pharmacokinet. 1997 May;32(5):345-56. doi: 10.2165/00003088-199732050-00001. No abstract available. PMID 9160169

DOCUMENTS (1):
  • Informed Consent Form (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02850900/ICF_000.pdf